CLINICAL TRIAL: NCT03026556
Title: Safety and Effectiveness Study Comparing Dabigatran, Rivaroxaban & Apixaban in Non-valvular Atrial Fibrillation Patients Enrolled in the US Department of Defense Military Health System
Brief Title: The Comparative Safety and Effectiveness of Dabigatran, Versus Rivaroxaban, and Apixaban Utilized in the Department of Defense Non-Valvular Atrial Fibrillation Patient Population: A Retrospective Database Analysis
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Health ResearchTx, LLC (HRTX) (Unknown); inVentiv Health Clinical (iVH) (Unknown); United States Department of Defense (DOD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1160-0274
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dabigatran vs. Rivaroxaban: OAC treatment naïve NVAF patients with at least one prescription claim for dabigatran, rivaroxaban (new oral anticoagulant or NOAC).
  Interventions: Drug: Dabigatran vs. Rivaroxaban
- Dabigatran vs. Apixaban: OAC treatment naïve NVAF patients with at least one prescription claim for dabigatran, or apixaban (new oral anticoagulant or NOAC).
  Interventions: Drug: Dabigatran vs. Apixaban

INTERVENTIONS:
Drug: Dabigatran vs. Rivaroxaban — observed for 6 years
  Groups: Dabigatran vs. Rivaroxaban
Drug: Dabigatran vs. Apixaban — Observed for 6 years
  Groups: Dabigatran vs. Apixaban

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of newly initiated dabigatran among patients diagnosed with non valvular atrial fibrillation (NVAF) in comparison to newly initiated rivaroxaban users and newly initiated apixaban users

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ on index date
* Patients must have been prescribed either dabigatran, rivaroxaban, or apixaban identified by pharmacy claim during the study period. The first dispensing date of either study drug will be defined as the index date;
* Patients must be treatment naïve from all OAC use prior to the first NOAC prescription, during study period.
* Patients must have at least 12 months of continuous eligibility prior to the index date;
* Patients must have at least one diagnosis code of atrial fibrillation, defined as International Classification of Diseases (ICD)-9-CM diagnosis of 427.31 or ICD-10-CM diagnosis of I48.0, I48.1, I48.2, I48.91 on the index date or during the pre-index period.

Exclusion Criteria:

Less than 12 months of continuous eligibility in the pre-index period Any claim for OAC drug (oral use only) in the pre-index period Diagnosis of hyperthyroidism during the pre-index period

Having at least one claim for alternative indications; orthopedic procedures, Venous thromboembolism (VTE) (includes deep vein thrombosis (DVT ) & PE)) and the index NOAC prescription at the same time, or, the alternative indication for anticoagulant occurring within 3 months prior to index date in pre-period Having at least one claim with any of the following diagnoses or procedure codes in order to exclude patients with "transient" causes of Afib (3 months prior to index date in pre-period):

* Cardiac surgery
* Pericarditis
* Myocarditis Having at least one medical claim with any of the following diagnoses or procedures codes in order to exclude patients with "valvular" Afib (pre-period):
* Mitral stenosis
* Mitral stenosis with insufficiency
* Mitral valve stenosis and aortic valve stenosis
* Mitral valve stenosis and aortic valve insufficiency
* Diseases of other endocardial structures
* Other and unspecified rheumatic heart diseases
* Open heart valvuloplasty without replacement
* Open and other replacement of unspecified heart valve
* Open and other replacement of aortic valve
* Open and other replacement of mitral valve
* Open and other replacement of pulmonary valve
* Open and other replacement of tricuspid valve
* Heart valve replaced by transplant
* Heart valve replaced by a mechanical device/prosthesis
* Atrioventricular valve repair
* Aortic valve valvuloplasty
* Unlisted procedure, cardiac surgery
* Implantation of catheter-delivered prosthetic aortic heart valve; open thoracic approach
* Transthoracic cardiac exposure (e.g., sternotomy, thoracotomy, subxiphoid) for catheter-delivered aortic valve replacement; without cardiopulmonary bypass
* Transthoracic cardiac exposure (e.g., sternotomy, thoracotomy, subxiphoid) for catheter-delivered aortic valve replacement; with cardiopulmonary bypass
* Replacement, aortic valve, with cardiopulmonary bypass; with prosthetic valve other than homograft or stentless valve
* Valvuloplasty, mitral valve, with cardiopulmonary bypass
* Valvuloplasty, mitral valve, with cardiopulmonary bypass; with prosthetic ring
* Valvuloplasty, mitral valve, with cardiopulmonary bypass; radical reconstruction, with or without ring
* Replacement, mitral valve, with cardiopulmonary bypass
* Implantation of catheter-delivered prosthetic pulmonary valve, endovascular approach
* Replacement, pulmonary valve
* Valvectomy, tricuspid valve, with cardiopulmonary bypass
* Valvuloplasty, tricuspid valve; without ring insertion
* Valvuloplasty, tricuspid valve; with ring insertion
* Replacement, tricuspid valve, with cardiopulmonary bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NVAF patients, ≥18 years of age, enrolled within the DoD Military Health System, who have newly initiated dabigatran, rivaroxaban, or apixaban. Patients must be treatment naïve from OAC use prior to first (index) NOAC.
Sampling Method: Non-Probability Sample
Enrollment: 42534 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inventiv Health, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Non-interventional retrospective cohort study based on existing data with propensity score matching (PSM) in Non-valvular Atrial Fibrillation (NVAF) patients with new Non-Vitamin K antagonist oral anticoagulant (NOAC) use.
Pre-assignment Details: The study was a US retrospective database of the Department of Defense (DoD) beneficiary population. Data was extracted from July 1, 2010 to June 30, 2016. Thus there was no pre-assignment/screening details.
Groups:
- Dabigatran: Oral anticoagulant (OAC) treatment naïve NVAF patients with at least one Non-Vitamin K antagonist oral anticoagulant (NOAC) prescription claim for dabigatran .
- Rivaroxaban: OAC treatment naïve NVAF patients with at least one NOAC prescription claim for rivaroxaban .
- Apixaban: OAC treatment naïve NVAF patients with at least one NOAC prescription claim for apixaban .
Period: Overall Study
Arm/Group | Dabigatran | Rivaroxaban | Apixaban
Started | 12763 | 17177 | 12594
Completed | 12763 | 17177 | 12594
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The main analysis was on matched patients based on their baseline characteristics using the propensity score matching (PSM) for the two study cohorts (dabigatran vs rivaroxaban and dabigatran vs apixaban cohorts). Baseline measures were presented for overall treatment groups and matched populations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Rivaroxaban | Apixaban | Total
Number analyzed (Participants) | 12763 | 17177 | 12594 | 42534
Age, Customized [Mean (Standard Deviation); unit: Years] — Population: The main analysis was on matched patients based on their baseline characteristics using the propensity score matching (PSM) for the two study cohorts (dabigatran vs rivaroxaban and dabigatran vs apixaban cohorts). Baseline measures were presented for overall treatment groups and matched populations.
  Years
    Overall | 70.89 (10.03) | 71.28 (9.70) | 72.35 (8.93) | 71.48 (9.60)
    Dabigatran vs Rivaroxaban (matched pop): number analyzed (Participants) | 12763 | 12763 | 0 | 25526
    Dabigatran vs Rivaroxaban (matched pop) | 70.89 (10.03) | 70.92 (10.07) |  | 70.91 (10.05)
    Dabigatran vs Apixaban (matched pop): number analyzed (Participants) | 4802 | 0 | 4802 | 9604
    Dabigatran vs Apixaban (matched pop) | 70.15 (10.23) |  | 70.20 (10.02) | 70.18 (10.13)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The main analysis was on matched patients based on their baseline characteristics using the propensity score matching (PSM) for the two study cohorts (dabigatran vs rivaroxaban and dabigatran vs apixaban cohorts). Baseline measures were presented for overall treatment groups and matched populations.
  Participants
    Overall: Male | 7902 | 10389 | 7499 | 25790
    Overall: Female | 4861 | 6788 | 5095 | 16744
    Dabigatran vs Rivaroxaban (matched pop): number analyzed (Participants) | 12763 | 12763 | 0 | 25526
    Dabigatran vs Rivaroxaban (matched pop): Male | 7902 | 7839 |  | 15741
    Dabigatran vs Rivaroxaban (matched pop): Female | 4861 | 4924 |  | 9785
    Dabigatran vs Apixaban (matched pop): number analyzed (Participants) | 4802 | 0 | 4802 | 9604
    Dabigatran vs Apixaban (matched pop): Male | 3028 |  | 3039 | 6067
    Dabigatran vs Apixaban (matched pop): Female | 1774 |  | 1763 | 3537
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity information was not collected for this trial. Population: The main analysis was on matched patients based on their baseline characteristics using the propensity score matching (PSM) for the two study cohorts (dabigatran vs rivaroxaban and dabigatran vs apixaban cohorts). Baseline measures were presented for overall treatment groups and matched populations.
  Participants
    Overall: White | 3771 | 5388 | 3744 | 12903
    Overall: Black | 302 | 358 | 272 | 932
    Overall: Other/Unknown/Missing | 8690 | 11431 | 8578 | 28699
    Dabigatran vs Rivaroxaban (matched pop): number analyzed (Participants) | 12763 | 12763 | 0 | 25526
    Dabigatran vs Rivaroxaban (matched pop): White | 3771 | 3779 |  | 7550
    Dabigatran vs Rivaroxaban (matched pop): Black | 302 | 297 |  | 599
    Dabigatran vs Rivaroxaban (matched pop): Other/Unknown/Missing | 8690 | 8687 |  | 17377
    Dabigatran vs Apixaban (matched pop): number analyzed (Participants) | 4802 | 0 | 4802 | 9604
    Dabigatran vs Apixaban (matched pop): White | 1621 |  | 1622 | 3243
    Dabigatran vs Apixaban (matched pop): Black | 157 |  | 152 | 309
    Dabigatran vs Apixaban (matched pop): Other/Unknown/Missing | 3024 |  | 3028 | 6052

OUTCOME MEASURES:

1. Primary Outcome: Stroke Overall (Hemorrhagic, Ischemic, Uncertain)
Description: The event rate of overall stroke (hemorrhagic, ischemic, uncertain) in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Length of Follow-up: The post-index follow-up period began the day following the NOAC index date and ended on whichever of the following occurred earliest:
  1. The day of discontinuation of the index NOAC exposure;
  2. The day before a switch to an anticoagulant different from the index exposure;
  3. The day before a change in dose for the index NOAC;
  4. The end of continuous eligibility of a patient in the health plan (disenrollment);
  5. The end of the study observation period; or
  6. The date of death of the patient.
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: Based on Department of Defense (DoD) outpatient prescription dispensed data the two separate study cohorts dabigatran vs rivaroxaban cohort and dabigatran vs apixaban cohort were formed. In both cohorts, dabigatran patients were matched 1:1 to comparator patients based on their baseline characteristics using the propensity score matching (PSM).
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Groups:
- Dabigatran (Dabigatran vs Rivaroxaban): OAC treatment naïve NVAF patients with at least one NOAC prescription claim for dabigatran; 1:1 matching of dabigatran to rivaroxaban was based on their baseline characteristics using the propensity score matching (PSM).
- Rivaroxaban (Dabigatran vs Rivaroxaban): OAC treatment naïve NVAF patients with at least one NOAC prescription claim for rivaroxaban; 1:1 matching of dabigatran to rivaroxaban was based on their baseline characteristics using the propensity score matching (PSM).
- Dabigatran (Dabigatran vs Apixaban): OAC treatment naïve NVAF patients with at least one NOAC prescription claim for dabigatran; 1:1 matching of dabigatran to apixaban was based on their baseline characteristics using the propensity score matching (PSM).
- Apixaban (Dabigatran vs Apixaban): OAC treatment naïve NVAF patients with at least one NOAC prescription claim for apixaban; 1:1 matching of dabigatran to apixaban was based on their baseline characteristics using the propensity score matching (PSM).
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 0.52 [0.41 to 0.66] | 0.69 [0.56 to 0.84] | 0.46 [0.28 to 0.70] | 0.36 [0.21 to 0.58]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); Cox proportional-hazards regression analysis was used to compute Hazard ratios (HR) and corresponding 95% confidence intervals (CI); Test type: Other; p = 0.0844, Regression, Cox; Hazard Ratio (HR) = 0.766, 95% CI 2-sided [0.566 to 1.037]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4892, Regression, Cox; Hazard Ratio (HR) = 1.255, 95% CI 2-sided [0.659 to 2.390]

2. Primary Outcome: Overall Major Bleeding
Description: The event rate of overall Major bleeding (Hemorrhagic Stroke, Major Intracranial Bleeding and Major Extracranial Bleeding) in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first.
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: Based on Department of Defense (DoD) outpatient prescription dispensed data the two separate study cohorts dabigatran vs rivaroxaban cohort and dabigatran vs apixaban cohort were formed and matched 1: 1 based on their baseline characteristics using the propensity score matching (PSM).
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 1.82 [1.60 to 2.05] | 2.24 [2.00 to 2.49] | 1.69 [1.33 to 2.11] | 1.24 [0.94 to 1.60]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0182, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.696 to 0.967]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0702, Regression, Cox; Hazard Ratio (HR) = 1.374, 95% CI 2-sided [0.974 to 1.939]

3. Secondary Outcome: Ischemic Stroke
Description: The event rate of ischemic stroke in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 0.5 [0.39 to 0.62] | 0.54 [0.42 to 0.67] | 0.39 [0.23 to 0.62] | 0.36 [0.21 to 0.58]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6307, Regression, Cox; Hazard Ratio (HR) = 0.923, 95% CI 2-sided [0.667 to 1.278]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.8777, Regression, Cox; Hazard Ratio (HR) = 1.054, 95% CI 2-sided [0.540 to 2.055]

4. Secondary Outcome: Hemorrhagic Stroke
Description: The event rate of Hemorrhagic stroke in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first.
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 0.03 [0.01 to 0.08] | 0.16 [0.11 to 0.25] | 0.07 [0.01 to 0.19] | NA [NA to NA] — As there is no person with the event of interest in apixaban groups thus event rate and 95% CI is not calculated
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0023, Regression, Cox; Hazard Ratio (HR) = 0.223, 95% CI 2-sided [0.085 to 0.585]

5. Secondary Outcome: Major Intracranial Bleeding
Description: The event rate of major intracranial bleeding in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 0.27 [0.19 to 0.37] | 0.41 [0.31 to 0.53] | 0.24 [0.12 to 0.43] | 0.21 [0.10 to 0.39]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0406, Regression, Cox; Hazard Ratio (HR) = 0.654, 95% CI 2-sided [0.435 to 0.982]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.8124, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.469 to 2.630]

6. Secondary Outcome: Major Extracranial Bleeding
Description: The event rate of major extracranial bleeding (Major GI bleeding, Major urogenital bleeding and Major other bleeding) in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 1.55 [1.35 to 1.76] | 1.83 [1.62 to 2.07] | 1.44 [1.12 to 1.84] | 1.03 [0.76 to 1.36]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0901, Regression, Cox; Hazard Ratio (HR) = 0.856, 95% CI 2-sided [0.716 to 1.025]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0616, Regression, Cox; Hazard Ratio (HR) = 1.431, 95% CI 2-sided [0.983 to 2.083]

7. Secondary Outcome: Major GI Bleeding
Description: The event rate of major GI bleeding (Upper GI Bleeding and Lower GI Bleeding) in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 1.45 [1.26 to 1.66] | 1.66 [1.46 to 1.89] | 1.36 [1.04 to 1.74] | 0.92 [0.66 to 1.24]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2073, Regression, Cox; Hazard Ratio (HR) = 0.887, 95% CI 2-sided [0.736 to 1.069]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0417, Regression, Cox; Hazard Ratio (HR) = 1.504, 95% CI 2-sided [1.015 to 2.228]

8. Secondary Outcome: Major Urogenital Bleeding
Description: The event rate of major urogenital bleeding in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first.
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | NA [NA to NA] — As there is no person with the event of interest for dabigatran in dabigatran vs rivaroxaban thus the event rate, 95% CI and Hazard ratio is not reported for dabigatran. | 0.01 [0.00 to 0.04] | NA [NA to NA] — As there is no person with the event of interest for dabigatran in dabigatran vs apixaban groups and also for the apixaban thus the event rate, 95% CI and Hazard ratio is not reported for dabigatran and for apixaban. | NA [NA to NA] — As there is no person with the event of interest for dabigatran in dabigatran vs apixaban groups and also for the apixaban thus the event rate, 95% CI and Hazard ratio is not reported for dabigatran and for apixaban.

9. Secondary Outcome: Major Other Bleeding
Description: The event rate of major other bleeding in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 0.13 [0.08 to 0.20] | 0.18 [0.12 to 0.26] | 0.11 [0.04 to 0.25] | 0.13 [0.05 to 0.28]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2663, Regression, Cox; Hazard Ratio (HR) = 0.709, 95% CI 2-sided [0.387 to 1.299]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.8112, Regression, Cox; Hazard Ratio (HR) = 0.864, 95% CI 2-sided [0.261 to 2.863]

10. Secondary Outcome: Upper GI Bleeding
Description: The event rate of Upper GI Bleeding in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 0.41 [0.31 to 0.52] | 0.55 [0.44 to 0.69] | 0.37 [0.22 to 0.59] | 0.34 [0.19 to 0.55]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.1227, Regression, Cox; Hazard Ratio (HR) = 0.766, 95% CI 2-sided [0.546 to 1.075]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.7115, Regression, Cox; Hazard Ratio (HR) = 1.138, 95% CI 2-sided [0.573 to 2.260]

11. Secondary Outcome: Lower GI Bleeding
Description: The event rate of Lower GI Bleeding in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 1.08 [0.91 to 1.26] | 1.17 [1.00 to 1.36] | 0.98 [0.72 to 1.32] | 0.58 [0.38 to 0.84]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4727, Regression, Cox; Hazard Ratio (HR) = 0.923, 95% CI 2-sided [0.741 to 1.149]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0275, Regression, Cox; Hazard Ratio (HR) = 1.721, 95% CI 2-sided [1.062 to 2.790]

12. Secondary Outcome: TIA
Description: The event rate of transient ischemic attack (TIA) in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 0.26 [0.18 to 0.35] | 0.20 [0.13 to 0.29] | 0.28 [0.15 to 0.48] | 0.17 [0.07 to 0.34]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2309, Regression, Cox; Hazard Ratio (HR) = 1.346, 95% CI 2-sided [0.828 to 2.189]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.3333, Regression, Cox; Hazard Ratio (HR) = 1.557, 95% CI 2-sided [0.635 to 3.821]

13. Secondary Outcome: All-cause Mortality
Description: The event rate of all-cause mortality in patients matched on propensity scores without index year.
  Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort.
  Follow-up time was the time elapsed from the index date to the date of the outcome of interest, disenrollment, end of the observation period (available data), death, discontinuation of the NOAC, or switch to a different NOAC, whichever came first
Time Frame: Baseline (July 1, 2010) until end of the observation period (June 30, 2016), 6 Years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Event Rate in 100 person-years
Arm/Group | Dabigatran (Dabigatran vs Rivaroxaban) | Rivaroxaban (Dabigatran vs Rivaroxaban) | Dabigatran (Dabigatran vs Apixaban) | Apixaban (Dabigatran vs Apixaban)
Number analyzed (Participants) | 12763 | 12763 | 4802 | 4802
Event Rate in 100 person-years | 1.54 [1.35 to 1.75] | 1.37 [1.18 to 1.57] | 1.46 [1.13 to 1.85] | 1.25 [0.96 to 1.62]
Statistical Analysis 1: Comparison: Dabigatran (Dabigatran vs Rivaroxaban) vs Rivaroxaban (Dabigatran vs Rivaroxaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.9359, Regression, Cox; Hazard Ratio (HR) = 1.008, 95% CI 2-sided [0.829 to 1.226]
Statistical Analysis 2: Comparison: Dabigatran (Dabigatran vs Apixaban) vs Apixaban (Dabigatran vs Apixaban); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.8947, Regression, Cox; Hazard Ratio (HR) = 1.024, 95% CI 2-sided [0.716 to 1.465]

ADVERSE EVENTS:
Description: This is a retrospective observational study, in which all patient data were de-identified and analyzed in aggregate. Individual patient safety related information were not captured during this study. Thus, individual safety reporting (including adverse events reporting) was not applicable for this study.
Groups:
- Dabigatran: Oral anticoagulant (OAC) treatment naïve NVAF patients with at least one Non-Vitamin K antagonist oral anticoagulant (NOAC) prescription claim for dabigatran.
- Rivaroxaban: OAC treatment naïve NVAF patients with at least one NOAC prescription claim for rivaroxaban.
- Apixaban: OAC treatment naïve NVAF patients with at least one NOAC prescription claim for apixaban.
Arm/Group | Dabigatran | Rivaroxaban | Apixaban
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT03026556/Prot_SAP_000.pdf